CLINICAL TRIAL: NCT05581810
Title: Feasibility of Cognitive Behavioural Therapy for Functional Memory Symptoms After Concussion
Brief Title: Rehabilitation for Functional Memory Symptoms After Concussion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Harvard Medical School (HMS and HSDM) (Other)
Responsible Party: Principal Investigator, Noah Silverberg, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H22-00436
Record Dates: First submitted 2022-09-22; First posted 2022-10-17 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Mild Traumatic Brain Injury; Functional Neurological Disorder
Keywords: Concussion; Functional Cognitive Disorder
MeSH Terms: conditions — Brain Concussion; Conversion Disorder | interventions — Cognitive Behavioral Therapy; Cognitive Training

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants will be blinded to their group assignment and treatment arms, but not to the type of intervention they are receiving. It is not possible to blind study therapists, as they have to administer the therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Behavioural Therapy (CBT) (Experimental): 11 weekly sessions of cognitive behavioural therapy (CBT) delivered over videoconference
  Interventions: Behavioral: Cognitive Behavioural Therapy (CBT)
- Cognitive Rehabilitation (Active Comparator): 11 weekly sessions of traditional cognitive rehabilitation delivered over videoconference
  Interventions: Behavioral: Cognitive Rehabilitation

INTERVENTIONS:
Behavioral: Cognitive Behavioural Therapy (CBT) — Cognitive behavioural therapy for functional memory symptoms after concussion is delivered by a psychologist over 11 individual (1:1) secure videoconference sessions. The core active ingredients are 1) Behavioural experiments, which acts by phasing out compensatory strategies in order to increase normal memory use and 2) Cognitive reappraisal, which aids in re-interpreting memory lapses in order to reduce reactivity to them.
  Arms: Cognitive Behavioural Therapy (CBT)
Behavioral: Cognitive Rehabilitation — Training and practice with external memory aids/compensatory strategies, adapted from Shum et al. (2011). J Rehabil Med, 43(3):216-223.
  Arms: Cognitive Rehabilitation

SUMMARY:
This study aims to evaluate the feasibility of novel cognitive behavioural therapy (CBT)-based intervention designed to improve functional memory symptoms after concussion. Participants will be randomized to CBT or an attention-matched control intervention (cognitive rehabilitation). The primary outcomes for this trial are feasibility metrics, including recruitment, patient-perceived credibility of treatment, patient adherence to treatment, therapists' compliance with the treatment protocol, and retention.

DETAILED DESCRIPTION:
Background: Although objectively measurable memory impairments typically resolve within weeks after sustaining a concussion, many people continue to perceive memory problems one year later. There are no known effective treatments for this condition. A promising new approach may be to target psychological mechanisms that perpetuate excessively negative perceptions of memory ability.

Methods: A pilot randomized controlled trial to evaluate the feasibility of a new cognitive behavioural therapy (CBT)-based treatment program specifically designed to improve persistent memory complaints after concussion. The main inclusion criteria will be (i) concussion in the past 6 to 24 months, (ii) research diagnosis of Functional Cognitive Disorder. Participants will be randomized (1:1) into one of two groups: CBT or cognitive rehabilitation. Individuals in both groups will participate in 11 x 50-minute sessions delivered over Zoom videoconference, co-facilitated by clinical psychology graduate students under the supervision of a registered clinical psychologist.

Aims: To evaluate the feasibility and potential efficacy of CBT for functional memory symptoms after concussion.

Approach: Prespecified feasibility criteria on recruitment, patient-perceived credibility of treatment, patient adherence to treatment, therapists' compliance with the treatment protocol, and retention will determine the success of the pilot trial. The investigators further hypothesize that CBT will be associated with greater reductions in memory concern compared to the control intervention.

Implications: The results of this pilot study will inform a larger, more definitive clinical trial focused on testing efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years old
* Fluent in English
* Have regular access to the internet
* Sustained a concussion according to the World Health Organization Neurotrauma Task Force definition between 6 and 24 months ago
* Meet diagnostic criteria for Functional Cognitive Disorder

Exclusion Criteria:

* Performance validity test failure
* Unstable/serious medical condition (e.g., cancer, multiple sclerosis, etc.),
* Unstable severe/mental illness (e.g., schizophrenia requiring hospital admission in the past year)
* Probable alcohol or drug use disorder
* Taking a medication with a known side effect of memory impairment (e.g., benzodiazepines, opiates, or topiramate)
* Contraindication(s) for MRI

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-11-29 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Recruitment | Week 0
  >50% of eligible participants agree to enroll
Treatment credibility | Week 2
  >50% of enrolled participants rate the intervention as above midpoint on credibility
Patient adherence | Week 12
  >70% of participants attend at least 8 sessions
Therapists compliance | Week 12
  Therapists cover 95% of essential element content
Retention | Week 12
  >80% of randomized participants complete the primary outcome measure immediately post-intervention
Memory concern | Week 12
  Satisfaction subscale of the Multifactorial Memory Questionnaire [range=0-72; higher scores indicate greater satisfaction with memory]

SECONDARY OUTCOMES:
Avoidance | Week 12
  Fear-Avoidance of Memory Loss Scale [range=5-25; higher scores indicate greater fear and avoidance]
Reliance on others | Week 12
  Relative subscale of the Memory Compensation Questionnaire [range=0-115; higher scores indicate greater dependence on others to remember things]
Catastrophizing | Week 12
  Adapted Pain Catastrophizing Scale [range=0-52, higher scores indicate greater catastrophizing]
Patient Global Impression of Change | Week 12
  Single item rated on a scale of 1 (much worse) to 5 (much better) since the start of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Noah Silverberg, PhD, Principal Investigator — University of British Columbia
Locations (10):
- Canada (10):
  - Urgent and Primary Care Center: North Vancouver, North Vancouver, British Columbia
  - Lion's Gate Hosital, North Vancouver, British Columbia
  - Richmond Hospital, Richmond, British Columbia
  - Back in Motion (Post-Concussion Management Program), Surrey, British Columbia
  - Mount Saint Joseph's Hospital, Vancouver, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia
  - Lifemark (Post-Concussion Management Program), Vancouver, British Columbia
  - University of British Columbia Hospital, Vancouver, British Columbia
  - Urgent and Primary Care Center: City Center, Vancouver, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia

IPD SHARING:
Plan to Share IPD: Yes
Upon reasonable request
Supporting Information: Study Protocol, ICF
Time Frame: 12 months after publication
Access Criteria: Defined research question approved by the principal investigator

REFERENCES:
- [Result] Rioux M, Mamman R, Byworth MT, Panenka WJ, Howard AK, Perez DL, Schmidt J, Courchesne C, LeMoult J, Heran MK, Silverberg ND. Pilot feasibility randomised controlled trial of cognitive-behavioural therapy for functional cognitive disorder after concussion. BMJ Neurol Open. 2024 Oct 11;6(2):e000666. doi: 10.1136/bmjno-2024-000666. eCollection 2024. PMID 39410977